CLINICAL TRIAL: NCT06015815
Title: The Association of MicroRNA-21 And MicroRNA-155 Levels With Acute Side Effects In Patients With Stage III Non Small Lung Cancer With Definite Chemoradiotherapy
Brief Title: The Association of MicroRNA21-155 Levels With Acute Side Effects In Patients With Stage III NSCLC With Definitive CRT
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Esra Gümüştepe, doctor research assistant, Ankara University
Other Study IDs: SRC Project No: 19L0230007
Record Dates: First submitted 2023-08-17; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Cancer Stage III
Keywords: Non-Small Cell Lung Cancer; Radiotherapy; MicroRNA-21; MicroRNA-155; Acute Side Effect
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — miRNA-21 and miRNA 155 in exosomes were examined in material from peripheral blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stage III non-small cell lung cancer: A total of 21 patients with stage III NSCLC who received definitive CRT were prospectively evaluated. The expression levels of miRNA-21 and miRNA-155 in serum at the beginning and end of the treatment

SUMMARY:
The present investigation constitutes a prospective cohort study. The objectives encompass the assessment of miRNA expression levels in total exosomes derived from peripheral circulation tissues of stage III definite KRT NSCLC patients both at the beginning and conclusion of their treatment. Furthermore, an exploration is conducted into the potential correlation existing between alterations in miRNA levels and the incidence of acute treatment-related side effects.

DETAILED DESCRIPTION:
Categorical variables were illustrated using both percentage distributions and numerical counts, while continuous variables were characterized using the mean accompanied by the standard deviation, and the median accompanied by the minimum and maximum values. The assessment of the normality of continuous variables encompassed a combination of visual methods such as histograms and probability plots, along with analytical tests like the Kolmogorov-Smirnov and Shapiro-Wilk tests.

In instances where data exhibited a normal distribution, Student's t-test was utilized for comparing two groups. For non-normally distributed data, the Mann-Whitney U test was applied. The comparison of categorical variables between independent groups involved Chi-square and Fisher's exact tests. Changes within dependent groups were evaluated using the Wilcoxon test. When performing pairwise comparisons among three or more groups, p-values were calculated while employing Bonferroni correction.

For the statistical analysis of the research data, the Statistical Package for Social Sciences (SPSS) version 25.0 for Windows (SPSS Inc. Chicago, USA) was utilized. The significance level was set at p<0.05. Additionally, it is important to note that p-values falling within the range of 0.1 to 0.05 were considered indicative of a statistical trend in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* To be between 0-2 according to Eastern Cooperative Oncology Group (ECOG) performance status (PS).
* Patient with pathological diagnosis of NSCLC.
* Stage 3 Patient
* Patient with a definitive chemoradiotherapy (CRT) treatment plan.

Exclusion Criteria:

* Patient with second primary malignancy.
* History of previous radiotherapy to the thoracic region
* Patient with advanced cardiovascular disease.
* Patient with neurological or physical deficit.
* Patient with autoimmune disease

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligibility criteria for inclusion in the study were defined as follows: patients aged 18 years or older who are histologically diagnosed with NSCLC and are in stage 3 according to the 8th edition of the American Cancer Committee (AJCC) staging system and are scheduled to receive treatment. During the staging of the patients, all of them underwent thorax computer tomography, positron emissions tomography (PET), and endobronchial ultrasound (EBUS) biopsy and cranial magnetic resonance imaging (MRI).
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
To determine the relationship of miRNA levels with acute side effects of chemoradiotherapy | The participants will be followed for an average of six months, including the period from the beginning of the treatment until three months after the completion of the treatment.
  miRNA Expression Measurement: Peripheral blood samples were collected from patients in pre-treatment and post-treatment periods to gauge miRNA expression. Samples were stored under suitable conditions. miRNA-21 and miRNA-155 expression levels were quantified through qRT-PCR. Livak formula-based fold change calculations identified expression shifts from treatment start to end.
  Acute Side Effects Assessment:
  Acute effects were evaluated as per Cooperative Group Common Toxicity Criteria Acute Side Effects (CTCAE) v5.0. Patients were assessed weekly during treatment and at 1 and 3 months post-treatment, comprehensively analyzing acute effects during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Gümüştepe, M.D, Principal Investigator — Ankara University; Serap Akyürek, M.D, Study Director — Ankara University
Locations (1):
- Ankara University Medicine School Radiation Oncology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No